CLINICAL TRIAL: NCT00506961
Title: A Phase IV, Randomized, Open-label, Parallel-arm, Comparative and Forced- Titration Study to Compare the Efficacy and Safety of Rosuvastatin Versus Simvastatin in Patients With Type 2 DM and Dyslipidemia
Brief Title: Evaluate the Efficacy and Safety of Rosuvastatin Versus Simvastatin in Type 2 Diabetic Patients With Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AZ-RSV-RT-01
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias | interventions — Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 10 mg rosuvastatin for 4 weeks followed by 20 m rosuvastatin for another 8 weeks
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): 20 mg simvastatin for 4 weeks followed by 40 mg simvastatin for another 8 weeks
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg rosuvastatin for 4 weeks followed by rosuvastatin or another 12 weeks
  Other Names: crestor
  Arms: 1
Drug: Simvastatin — 20 mg simvastatin for 4 weeks followed by 40 mg simvastatin for another 8 weeks
  Other Names: zocor
  Arms: 2

SUMMARY:
This is a phase IV, randomized, open-label, parallel-arm, comparative and forced- titration study to compare the efficacy and safety of rosuvastatin versus simvastatin in patients with type 2 DM and dyslipidemia. When comparing the efficacy of rosuvastatin 20 mg with simvastatin 40 mg for the treatment of type 2 DM with dyslipidemia, rosuvastatin 20 mg is superior to simvastatin 40 mg in achieving the combined goal of LDL-C (<100 mg/dL) and non-HDL-C (<130 mg/dL).

DETAILED DESCRIPTION:
The duration of patient participation will be 18 weeks consisting of a 1-week screening period, a 5-week lead-in period, followed by a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between the ages of 20-75 years.
2. Female patients post menopausal, hysterectomized or if of childbearing potential using a reliable method of birth control.
3. Diagnosed with type 2 diabetes mellitus.
4. Fasting triglyceride ≧150 mg/dL ≦500 mg/dL or Non-HDL-C≧130,but≦200 mg/dL
5. Patients receiving stable antidiabetic treatment for 8 weeks before randomization (no change in the category of anti-diabetic agents, but the dose is adjustable).
6. All patients give written informed consent.

Exclusion Criteria:

1. A history of hypersensitivity to statins.
2. A history of rhabdomyolysis or hereditary muscle disorders.
3. Insulin-treated patients.
4. Patient with any conditions of acute or chronic pancreatitis.
5. Creatine kinase ≧3-fold upper limit of normal (ULN).
6. Patients with an estimated creatinine clearance (see note)≦30 ml/min or bilirubin ≧1.5-fold ULN, or chronic active hepatitis or liver function impairment (AST and ALT ≧3-fold ULN).
7. Overt proteinuria (repeat spot urine protein >300mg/dl by dipstick method).
8. Patients are taking cyclosporine.
9. A history of homozygous familial hypercholesterolemia or familial dysbetalipoproteinemia.
10. Patients with alcohol and drug abuse in past 3 years.
11. Serious or unstable medical or psychological conditions.
12. Hypothyroidism (TSH > 5 μIU/mL).
13. In the investigator's opinion, continuation in the study would be detrimental to the patient's well-being or might confound the clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients achieving the combined treatment goal of LDL-C < 100mg/dl and non-HDL-C < 130 mg/dl at week 12 with rosuvastatin treatment compared with simvastatin treatment | 12 weeks

SECONDARY OUTCOMES:
Achieving the combined treatment goal of LDL-C (<100 mg/dL) and non-HDL-C (130 mg/dL) at week 4; | 4 weeks
Percentage of patients achieving the LDL-C goal of <100 mg/dL at week 4 and week 12; | 12 weeks
Percentage of patients achieving the LDL-C goal of <70 mg/dL at Week;The mean percent change from baseline in lipid profile at week 4 and week 12; | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Wayne H Sheu, MD,phD, Principal Investigator — Taichung Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Wu TH, Lee IT, Ho LT, Sheu WH, Hwu CM. Combined lipid goal attainment in patients with type 2 diabetes and dyslipidemia: A head-to-head comparative trial of statins. J Chin Med Assoc. 2022 Aug 1;85(8):831-838. doi: 10.1097/JCMA.0000000000000765. Epub 2022 Jun 20. PMID 35727095